CLINICAL TRIAL: NCT03973710
Title: Role of Probiotics in the Prevention of Hypertension
Brief Title: Effect of Probiotics on Blood Pressure Management
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough intervention materials can be provided
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Min Xia, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ProHealth-2
Record Dates: First submitted 2019-06-03; First posted 2019-06-04 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Hypertension
Keywords: Probiotics; Prevention; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, investigators and care providers at the scene are all blinded to the allocation of treatment group. Data collected will be analyzed by another investigator who is blinded to the study design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics group (Experimental): Participants will be given capsules containing Lactobacillus paracasei once daily for 12 weeks followed by comprehensive physical and clinical examinations.
  Interventions: Dietary Supplement: Lactobacillus paracasei dietary supplement
- Placebo group (Placebo Comparator): Participants will be given capsules containing microcrystalline cellulose once daily for 12 weeks followed by comprehensive physical and clinical examinations.
  Interventions: Dietary Supplement: Placebo controls

INTERVENTIONS:
Dietary Supplement: Lactobacillus paracasei dietary supplement — a commercial probiotic dietary supplement
  Arms: Probiotics group
Dietary Supplement: Placebo controls — placebo with a similar appearance to probiotics supplement
  Arms: Placebo group

SUMMARY:
Dysbiosis of gut microbiota has been reported to be involved in the development and progression of hypertension in both humans and animal models. Probiotics have been reported to have ameliorative effects in murine models. However, whether probiotics could help alleviate hypertension in adults remain obscure.

DETAILED DESCRIPTION:
Probiotics are live microorganisms that have been associated with multiple health benefits. However, its protective role in adults has long been controversial. This study aims to examine the effect of 12-week probiotics supplementation on the prevention of hypertension in Chinese adults. By understanding the mechanisms by which probiotics exert this beneficial effects, we can better control the rising prevalence of hypertension, which is a major risk factor for cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects include men and women 18 to 75 years of age with pre-hypertension who has a systemic blood between 120 and 139 mmHg and/ or a diastolic blood pressure between 80 and 80 mmHg;
* Absence of any diet, dietary supplement and medications that might interfere with blood pressure and gut microbiota, especially antibiotics and probiotics.

Exclusion Criteria:

* Any other systemic, metabolic and cardiovascular or cerebrovascular diseases;
* Type 1 diabetes, type 2 diabetes treated with insulin or other medications;
* Acute illness or current evidence of acute or chronic inflammatory or infective diseases;
* Participation in any diet or lifestyle program more than 2 times per week in the latest 3 months prior to recruitment;
* Mental illness rendering them unable to understand the nature, scope, and possible consequences of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-03 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
changes of systolic blood pressure | baseline, 4 weeks, 8 weeks and 12 weeks
  changes of systolic blood pressure
changes of diastolic blood pressure | baseline, 4 weeks, 8 weeks and 12 weeks
  changes of diastolic blood pressure
changes of gut microbiota | baseline, 4 weeks, 8 weeks and 12 weeks
  changes of gut microbiota by metagenomics

SECONDARY OUTCOMES:
changes of pulse wave velocity | baseline and after 12-week intervention
  changes of pulse wave velocity
changes of ankle brachial index | baseline and after 12-week intervention
  changes of ankle brachial index
changes of microbial metabolite | baseline and after 12-week intervention
  changes of microbial metabolite by untargeted metabolomics

CONTACTS AND LOCATIONS:
Overall Officials: Min Xia, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Nutrition and Food Hygiene, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No